CLINICAL TRIAL: NCT00512538
Title: A Randomized, Open-Label, Multi-Center Study to Compare the Safety and Efficacy of Apligraf Versus Standard Therapy (i.e., Saline Moistened Dressing Regimen) in the Treatment of Diabetic (Primarily Neuropathic) Foot Ulcers
Brief Title: Apligraf Versus Standard Therapy in the Treatment of Diabetic Foot Ulcers
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interruption of business relations between Study Sponsor and Device Manufacturer
Sponsor: Organogenesis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CGS0769 B304
Record Dates: First submitted 2007-08-03; First posted 2007-08-07 (Estimated); Last update posted 2007-08-07 (Estimated); Status verified 2007-08

CONDITIONS: Diabetic Foot
Keywords: Diabetic foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Bi-layered cell therapy (Apligraf)

SUMMARY:
The purpose of this study is to determine the ability of Apligraf to improve the time to and incidence of complete wound closure of diabetic foot ulcers, as compared to diabetic foot ulcers treated with standard therapy.

DETAILED DESCRIPTION:
Ulceration of the diabetic foot is a result of multiple problems including repetitive stress on a neuropathic or insensate area that is often associated with an underlying bony prominence. By healing diabetic foot ulcers quickly the risks of infection, osteomyelitis (infeciton of the bone) and limb loss can be reduced.

This study will evaluate the ability of Apligraf to heal diabetic foot ulcers that have been present for at least 2 weeks and are between 1 - 16 cm2 in area. Patients will be randomized to either (50:50 chance) treatment with Apligraf or a saline moistened dressing regimen (standard therapy). All patients will receive standard cares for the ulcers which includes debridement, orthotics and off-loading throughout the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* diabetic ulcer of primarily neuropathic origin on the plantar region of the forefoot
* ulcer extending through the dermis but without sinus tract, tendon, capsule or bone exposure
* ulcer present for at least 2 weeks and measuring 1- 16 cm2
* diminished sensesation on target extremity/foot
* ulcer is not infected
* Type 1 or 2 diabetes with adequate glycemic control
* Adequate vascular supply to the target extremity

Exclusion Criteria:

* Charcot foot
* Non-neuropathic ulcers
* Skin cancer within or adjacent to the target ulcer
* Osteomyelitis or an infected ulcer
* Clinically significant medical condition that would impair wound healing
* Females who are pregnant
* Received within 4 weeks of study entry systemic corticosteriods, immunosuppresive agents, radiation therapy or chemotherapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2000-10; Study Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
Time to complete wound healing (full epithelialization with no drainage) | through 12 weeks

SECONDARY OUTCOMES:
Incidence of complete healing | at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Edmonds, MD, Principal Investigator — Diabetic Foot Clinic, Kings College Hospital, London UK